CLINICAL TRIAL: NCT06332638
Title: Phase 1 Clinical Trial to Explore Pharmacokinetics, Pharmacodynamics and Safety of Tegoprazan 12.5 mg After Oral Administration in Healthy Subjects
Brief Title: PK, PD and Safety of Tegoprazan 12.5 mg After Oral Administration in Healthy Subjects
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN_APA_124
Record Dates: First submitted 2024-02-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — tegoprazan; Famotidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Tegoprazan 12.5mg
  Interventions: Drug: Tegoprazan 12.5mg
- Group B (Active Comparator): Tegoprazan 25mg
  Interventions: Drug: Tegoprazan 25mg
- Group C (Active Comparator): Famotidine 20mg
  Interventions: Drug: Famotidine 20mg

INTERVENTIONS:
Drug: Tegoprazan 12.5mg — Oral administration of one tablet of Tegoprazan 12.5mg twice daily for 14 days.
  Other Names: Tegoprazan Tab. 12.5mg
  Arms: Group A
Drug: Tegoprazan 25mg — Oral administration of one tablet of Tegoprazan 25mg once daily for 14 days.
  Other Names: K-CAB Tab. 25mg
  Arms: Group B
Drug: Famotidine 20mg — Oral administration of one tablet of Famotidine 20mg twice daily for 14 days.
  Other Names: Gaster Tab. 20 mg Dong-A
  Arms: Group C

SUMMARY:
The primary objective of this study is to explore pharmacokinetics, pharmacodynamics, and safety of tegoprazan 12.5 mg in healthy subjects when orally administered as a single dose or as multiple doses twice daily.

DETAILED DESCRIPTION:
The secondary objectives of this study are

* To compare pharmacokinetics and pharmacodynamics of tegoprazan 12.5 mg in healthy subjects between oral multiple-dose administration twice daily for 1 day and oral single-dose administration.
* To evaluate pharmacokinetics and pharmacodynamics of tegoprazan 12.5 mg administered orally twice daily for 14 days in healthy subjects in comparison with tegoprazan 25 mg administered orally once daily for 14 days in healthy subjects.
* To evaluate pharmacodynamics of tegoprazan 12.5 mg administered orally twice daily for 14 days or tegoprazan 25 mg administered orally once daily for 14 days in healthy subjects in comparison with famotidine 20 mg administered orally twice daily for 14 days in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged ≥ 19 years to ≤ 45 years at the time of screening testing
2. Body mass index (BMI) ≥ 18.5 kg/m2 to ≤ 28.0 kg/m2 (BMI = weight (kg) / height (m)2)
3. Those who have been fully informed of study purpose and procedures, properties of the investigational products(IPs), etc. and have voluntarily decide to participate in this study and signed an informed consent form (ICF), prior to participation in the study

Exclusion Criteria:

1. Medical history

   1. Previous history or presence of clinically significant hepatic, renal, gastrointestinal, respiratory, musculoskeletal, endocrine, neuropsychiatric, hemato-oncologic, urinary and cardiovascular (including cardiac arrhythmia) disorders in the judgment of the investigator
   2. Previous history of gastrointestinal diseases (e.g., gastritis, gastrospasm, gastroesophageal reflux disease (GERD), Crohn's disease, ulcers, etc.) or abdominal surgery (excluding simple appendectomy or hernia surgery) which may affect drug absorption in the judgment of the investigator
   3. Presence of anatomical disorders that make it difficult to insert and maintain a catheter for intragastric pH measurement, or expected intolerance to catheterization for intragastric pH measurement
   4. Hereditary problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
2. Clinical laboratory tests and electrocardiogram (ECG)

   1. AST or ALT value ≥ 1.5 x upper limit of normal (ULN) as a result of clinical laboratory testing at screening
   2. Total bilirubin value ≥ 2.0 x upper limit of normal (ULN) as a result of clinical laboratory testing at screening
   3. eGFR value calculated using the CKD-EPI formula < 80 mL/min as a result of clinical laboratory testing at screening
   4. Any clinically significant abnormality as a result of ECG at screening
   5. Positive test result for H. pylori at screening
3. Allergies and drug abuse

   1. History of hypersensitivity to the IPs, components of the IPs, and other drugs (benzimidazoles, H2 receptor antagonists, aspirin, antibiotics, etc.)
   2. Previous history of drug abuse or positive drug screening test result
4. Prohibited concomitant medications/diets

   1. Consumption of medicines (including herbal medicines) or abnormal diets (e.g., at least 1L/day of grapefruit juice, much garlic, broccoli, kale, etc.) which may affect the absorption, distribution, metabolism, and excretion of the IP within 28 days before the screening visit
   2. Administration of the drugs affecting gastric pH within 14 days before the screening visit (including potassium-competitive acid blockers, proton pump inhibitors, H2-receptor antagonists, and antacids) or administration of ethical-the-counter (ETC) drugs, any over-the-counter (OTC) drugs, vitamins, etc. within 10 days before the screening visit
   3. Administration of another IP by participating in another clinical trial within 6 months prior to the screening visit (but those who are not administered the IP can participate in this study)
5. Blood donation and transfusion

   1. Whole blood donation within 60 days before the screening visit
   2. Blood component donation or transfusion within 30 days before the screening visit
6. Pregnancy, breastfeeding, and non-use of contraceptives

   1. Pregnant women, women who tested positive for pregnancy, or breastfeeding women
   2. Failure to use medically recognized and proper double contraceptive methods or medically acceptable contraceptive methods (intrauterine device showing a demonstrated pregnancy failure rate, combined use of physical barrier method and spermicide, vasectomy, salpingectomy/tubal ligation, hysterectomy, etc.) in the subject or his/her spouse or partner from the date of screening visit until 30 days after the last dose of the IP
7. Others

   1. Mean alcohol intake exceeding 30 g/day per week for recent 4 weeks before the screening visit or positive alcohol breath test result
   2. Mean number of smoked cigarettes exceeding 10 cigarettes/day per week for recent 4 weeks before the screening visit
   3. Mean caffeine intake exceeding 400 mg/day per week for recent 4 weeks before the screening visit
   4. Presence of clinically significant findings that make the subject ineligible for this study in the judgment of the investigator

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Cmax of tegoprazan and tegoprazan's metabolite M1 | Pre-dose(0 hour) up to 24 hours on Day 1
  Pharmacokinetic evaluation (Day 1)
AUC0-t of tegoprazan and tegoprazan's metabolite M1 | Pre-dose(0 hour) up to 24 hours on Day 1
  Pharmacokinetic evaluation (Day 1)
AUC0-∞ of tegoprazan and tegoprazan's metabolite M1 | Pre-dose(0 hour) up to 24 hours on Day 1
  Pharmacokinetic evaluation (Day 1)
Tmax of tegoprazan and tegoprazan's metabolite M1 | Pre-dose(0 hour) up to 24 hours on Day 1
  Pharmacokinetic evaluation (Day 1)
t1/2β of tegoprazan and tegoprazan's metabolite M1 | Pre-dose(0 hour) up to 24 hours on Day 1
  Pharmacokinetic evaluation (Day 1)
CL/F of tegoprazan | Pre-dose(0 hour) up to 24 hours on Day 1
  Pharmacokinetic evaluation (Day 1)
Vd/F of tegoprazan | Pre-dose(0 hour) up to 24 hours on Day 1
  Pharmacokinetic evaluation (Day 1)
Css,max of tegoprazan and tegoprazan's metabolite M1 | Pre-dose(morning) (-12, 0 hour) up to 24 hours on Day 14
  Pharmacokinetic evaluation (Day 14)
Css,min of tegoprazan and tegoprazan's metabolite M1 | Pre-dose(morning)(-12, 0 hour) up to 24 hours on Day 14
  Pharmacokinetic evaluation (Day 14)
Css,avg of tegoprazan and tegoprazan's metabolite M1 | Pre-dose(morning)(-12, 0 hour) up to 24 hours on Day 14
  Pharmacokinetic evaluation (Day 14)
AUCtau,ss of tegoprazan and tegoprazan's metabolite M1 | Pre-dose(morning)(-12, 0 hour) up to 24 hours on Day 14
  Pharmacokinetic evaluation (Day 14)
Tmax,ss of tegoprazan and tegoprazan's metabolite M1 | Pre-dose(morning)(-12, 0 hour) up to 24 hours on Day 14
  Pharmacokinetic evaluation (Day 14)
t1/2β,ss of tegoprazan and tegoprazan's metabolite M1 | Pre-dose(morning)(-12, 0 hour) up to 24 hours on Day 14
  Pharmacokinetic evaluation (Day 14)
CLss/F of tegoprazan | Pre-dose(morning)(-12, 0 hour) up to 24 hours on Day 14
  Pharmacokinetic evaluation (Day 14)
Vdss/F of tegoprazan | Pre-dose(morning)(-12, 0 hour) up to 24 hours on Day 14
  Pharmacokinetic evaluation (Day 14)
Accumulation index of tegoprazan | Pre-dose(morning)(-12, 0 hour) up to 24 hours on Day 14
  Pharmacokinetic evaluation (Day 14)
Fluctuation of tegoprazan | Pre-dose(morning)(-12, 0 hour) up to 24 hours on Day 14
  Pharmacokinetic evaluation (Day 14)

SECONDARY OUTCOMES:
24-hour, daytime and nighttime mean pH | 24 hours on Day -1, Day 1, Day 7, and Day 14
  Pharmacodynamic evaluation
24-hour, daytime and nighttime median pH | 24 hours on Day -1, Day 1, Day 7, and Day 14
  Pharmacodynamic evaluation
24-hour, daytime and nighttime TpH>3(%) | 24 hours on Day -1, Day 1, Day 7, and Day 14
  Pharmacodynamic evaluation
24-hour, daytime and nighttime TpH>4(%) | 24 hours on Day -1, Day 1, Day 7, and Day 14
  Pharmacodynamic evaluation
24-hour, daytime and nighttime Δ TpH>3(%) | 24 hours on Day -1, Day 1, Day 7, and Day 14
  Pharmacodynamic evaluation
24-hour, daytime and nighttime Δ TpH>4(%) | 24 hours on Day -1, Day 1, Day 7, and Day 14
  Pharmacodynamic evaluation
24-hour, daytime and nighttime Δ mean pH | 24 hours on Day -1, Day 1, Day 7, and Day 14
  Pharmacodynamic evaluation
24-hour, daytime and nighttime Δ median pH | 24 hours on Day -1, Day 1, Day 7, and Day 14
  Pharmacodynamic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Jong Lyul Ghim, MD, PhD, Principal Investigator — Department of Clinical Pharmacology, Inje University Busan Paik Hospital
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea